CLINICAL TRIAL: NCT01196832
Title: Role of Fibrocytes in the Bronchial Remodeling of Chronic Obstructive Pulmonary Disease
Brief Title: Role of Fibrocytes in Chronic Obstructive Pulmonary Disease
Acronym: FIREBROB
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/05
Record Dates: First submitted 2010-06-01; First posted 2010-09-09 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic obstructive pulmonary disease patients: COPD patients with exacerbation will be recruited during hospitalization in Intensive care unit or as outpatients in the clinical investigation centre of the CHU de Bordeaux.
  Inclusion visit: blood sample for fibrocytes analysis. Second visit 2 months ± 7 days after the exacerbation: clinical and functional evaluation (plethysmography, TLCO, arterial gaz), blood sample for fibrocytes analysis.
  Interventions: Procedure: blood sample; Procedure: Clinical and functional evaluation
- Control group: Subjects without any history of lung disease and with normal lung function testing
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — blood sample for fibrocytes analysis
Procedure: Clinical and functional evaluation — Plethysmography, Carbon monoxide capacity of transfer , arterial gaz
  Groups: Chronic obstructive pulmonary disease patients

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a frequent airway disease characterized by both bronchial inflammation and remodelling.

Bronchial mucosa is infiltrated by macrophages, neutrophils and lymphocytes. In addition, the number of eosinophils can be also increased during exacerbation.

Airway remodelling is an abnormal tissue repair following bronchial inflammation, which contributes to none reversible pathological features, such as bronchial and peri-bronchial fibrosis. It also influences the prognosis of COPD and its mechanisms remain largely unknown. The role of fibrocytes has been demonstrated in the pathophysiology of asthma, lung fibrosis or pulmonary hypertension. However, the recruitment of blood fibrocytes and their involvement in COPD airway remodelling remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients: diagnostic of Chronic obstructive pulmonary disease (COPD) exacerbation.
* Control group: subjects without any history of lung disease and with normal lung function testing. Subjects will be separated in 2 sub-groups according to smoking history (Never smokers, smokers (former or current) and paired to patients according to age and sex.
* Written informed consent

Exclusion Criteria:

* Subject without any social security or health insurance
* Asthma, lung fibrosis or idiopathic pulmonary hypertension
* Chronic viral infections (hepatitis, HIV)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female aged more than 40 years
  * Chronic obstructive pulmonary disease (CODP) patients recruited during hospitalization in Intensive care unit or as outpatients in the clinical investigation centre of the CHU de Bordeaux.
  * Control group: subjects without any history of lung disease and with normal lung function testing recruited following a normal lung function testing in the clinical investigation centre of the CHU de Bordeaux.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Number of circulating blood fibrocytes | Day 1
  Sampling of blood in Chronic obstructive pulmonary disease patients
Number of circulating blood fibrocytes | 2 months
  Sampling of blood in Chronic obstructive pulmonary disease patients

SECONDARY OUTCOMES:
Characterization of fibrocytes | Day 1 and at 2 months
  Sampling of blood
Differenciation of blood fibrocytes | Day 1 and at 2 months
  Sampling of blood
Chemotactism of blood fibrocytes | Day 1 and at 2 months
  Sampling of blood
Number of exacerbation | 12 months after V2
Mortality | 12 months after V2
Annual decline of ventilatory function | 12 months after V2

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BERGER, PUPH, Principal Investigator — University Hospital Bordeaux (France)
Locations (1):
- CHU de Bordeaux, Pessac, France

REFERENCES:
- [Derived] Dupin I, Allard B, Ozier A, Maurat E, Ousova O, Delbrel E, Trian T, Bui HN, Dromer C, Guisset O, Blanchard E, Hilbert G, Vargas F, Thumerel M, Marthan R, Girodet PO, Berger P. Blood fibrocytes are recruited during acute exacerbations of chronic obstructive pulmonary disease through a CXCR4-dependent pathway. J Allergy Clin Immunol. 2016 Apr;137(4):1036-1042.e7. doi: 10.1016/j.jaci.2015.08.043. Epub 2015 Oct 23. PMID 26602164